

## **Croydon University Hospital**

530 London Road Croydon CR7 7YE

Switchboard Tel: (020) 8401 3000

## **Informed Consent Form**

Study Number:

Women & Children's Directorate

Direct Line Tel: (020) 8401-3145 Direct Fax: (020) 8401-3681 Email: Ranee.Thakar@mayday.nhs.uk

CIVIL - Copper Impact on Venous Insufficiency and Lipodermatosclerosis

| Please | sian | the | box | with | initia | ls |
|--------|------|-----|-----|------|--------|----|

| 1. | I confirm that I have read an sheet, dated 17/03/2015, for the opportunity to ask questi | | |
|---|---|---|---|
| 2. | I understand that my particip<br>free to withdraw at any time<br>without my medical care or I | | |
| 3. | I understand that sections of<br>at by responsible individuals<br>my taking part in research. I<br>to have access to my record | | |
| 4. | I understand that photograph<br>after 2, 4 and 8 weeks. I give<br>my legs. | | |
| 5. | I consent for my GP to be in study. | | |
| 6. | I agree to take part in this st | udy. | |
| Name | of patient | Date | Signature |
| Name | of researcher | Date | Signature |

CIVIL study (15/LO/0974)

Version 1
17-03-2015